CLINICAL TRIAL: NCT00005589
Title: Randomized Study of Rituximab (Mabthera) in Patients With Relapsed Follicular Lymphoma Prior to High-Dose Therapy as In Vivo Purging and to Maintain Remission Following High-Dose Therapy
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation With or Without Rituximab in Treating Patients With Relapsed Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EBMT Solid Tumors Working Party (Other)
Collaborators: Lymphoma Trials Office (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067665; EBMT-EBMTLYM1; BNLI-EBMT-EBMTLYM1; EU-99050
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-03

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — Filgrastim; Rituximab; Carmustine; Cyclophosphamide; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Biological: rituximab
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: etoposide
Drug: melphalan
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known if combination chemotherapy plus peripheral stem cell transplantation is more effective with or without rituximab for non-Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy and peripheral stem cell transplantation together with rituximab to see how well it works compared to combination chemotherapy and peripheral stem cell transplantation alone in treating patients with relapsed non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effects of in vivo rituximab purging and maintenance on progression-free survival in patients with relapsed or resistant follicular non-Hodgkin's lymphoma undergoing high-dose chemotherapy.
* Determine the effects of this regimen on response rate and overall survival in this patient population.
* Determine the effects of in vivo purging with rituximab on molecular remission rates in the hematopoietic product and the patients.
* Determine the safety of rituximab in the transplant setting.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to type of remission (complete vs good partial) and which remission (second vs third). Patients are randomized to one of four treatment arms.

All patients receive induction chemotherapy comprising cyclophosphamide IV over 3-4 hours on day 0 or a standard induction chemotherapy regimen. Filgrastim (G-CSF) is administered subcutaneously daily beginning on day 1.

Patients are then randomized to receive either in vivo rituximab purging or no purging following restaging after completion of induction. For those patients receiving purging (arms I and II), rituximab is administered IV once weekly for 4 weeks.

Peripheral blood stem cells (PBSC) are collected between days 8 and 12 post induction chemotherapy. Within 4 weeks of PBSC collection, patients receive carmustine IV over 2 hours on day -6, etoposide IV over 2 hours on days -5 to -2, cytarabine IV over 5 minutes twice daily on days -5 to -2, and melphalan IV over 10-15 minutes on day -1. (Alternatively, high dose cyclophosphamide and total body irradiation beginning 2-4 weeks after cyclophosphamide or standard induction chemotherapy priming is also allowed.) PBSC are reinfused on day 0.

Patients are further randomized to receive either rituximab maintenance or observation only. For those patients receiving maintenance (arms I and III), rituximab is administered IV once every 2 months for 4 doses beginning 30 days after PBSC reinfusion.

Patients are followed at 30 days, 3, 6, 9, and 12 months after PBSC transplant, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 460 patients (115 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Relapsed or resistant follicular non-Hodgkin's lymphoma (NHL)

  * No evidence of transformation to high grade or diffuse large B-cell NHL
* CD20 positive with no evidence of transformation
* Achievement of complete remission (CR) or very good partial remission (VGPR) following reinduction chemotherapy with any standard regimen

  * Includes patients who fail to respond to first-line chemotherapy but who achieve CR or VGPR after proceeding directly to second-line chemotherapy
* Platelet count greater than 100,000/mm^3 after induction chemotherapy and before randomization
* No CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-1

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Bilirubin normal
* ALT no greater than 2 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2 times ULN
* Hepatitis B negative
* Hepatitis C negative

Renal:

* Creatinine no greater than 2 times ULN
* BUN no greater than 2 times ULN

Cardiovascular:

* No inadequate cardiac function

Pulmonary:

* No inadequate pulmonary function

Other:

* Not pregnant or nursing
* HIV negative
* No other uncontrolled serious medical conditions
* No other malignancy within the past 5 years except nonmelanoma skin tumors or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 12 months since prior CD20 therapy, including rituximab
* No prior peripheral blood stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* No more than 3 prior chemotherapy regimens for NHL

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to greater than 30% of bone marrow

Surgery:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 1999-10; Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time to disease progression

SECONDARY OUTCOMES:
Response rate and survival
Molecular remission rates
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Pettengell, MD, Study Chair — St George's, University of London; David C. Linch, Study Chair — Middlesex Hospital
Locations (131):
- Australia (8):
  - Sydney Cancer Centre at Royal Prince Alfred Hospital, Sydney, New South Wales
  - Westmead Institute for Cancer Research at Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Royal Adelaide Hospital Cancer Centre, Adelaide, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Allgemeines Krankenhaus - Universitatskliniken, Vienna, Austria
- Belgium (8):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Academisch Ziekenhuis der Vrije Universiteit Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - U.Z. Gasthuisberg, Leuven
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
  - H. Hartziekenhuis - Roeselaere., Roeselaere
- Canada (2):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
- University Hospital Kralovske Vinohr, Prague, Czechia
- Denmark (3):
  - Aalborg Hospital, Aalborg
  - Rigshospitalet - Copenhagen University Hospital, Copenhagen
  - Odense University Hospital, Odense
- France (15):
  - Centre Hospitalier Regional et Universitaire d'Angers, Angers
  - Polyclinique Du Parc, Caen
  - Centre Regional Francois Baclesse, Caen
  - CHU de Grenoble - Hopital de la Tronche, Grenoble
  - Centre Leon Berard, Lyon
  - Polyclinique Saint Jean, Melun
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CHR Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - CHU Pitie-Salpetriere, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (9):
  - Klinikum Augsburg, Augsburg
  - DIAKO Ev. Diakonie Krankenhaus gGmbH, Bremen
  - Universitaetsklinikum Goettingen, Göttingen
  - Asklepios Klinik St. Georg, Hamburg
  - Medical University Hospital Homburg, Homburg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Klinikum Oldenburg, Oldenburg
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
- Chaim Sheba Medical Center, Tel Litwinsky, Israel
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Canterbury Health Laboratories, Christchurch
  - Waikato Hospital, Hamilton
- Poland (2):
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
  - K. Dluski Hospital-Medical Academy, Wroclaw
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- Spain (34):
  - Hospital Juan Canalejo, A Coruña
  - Hospital General - Alicante, Alicante
  - Hospital de Cruces, Barakaldo Bilbao
  - Centro Medico Teknon, Barcelona
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Puerta Del Mar, Cadiz
  - Hospital General de Castellon, Castellon
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Virgen de la Arrixaca, El Palmar
  - Hospital de Galdakao, Galdakao Vizcaya
  - Hospital Virgen de las Nieves, Granada
  - Hospital Cuidad de Jaen, Jaén
  - Hospital de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital de la Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Getafe, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Son Dureta, Palma de Mallorca
  - Hospital Virgen de la Vega, Salamanca
  - University Hospital - Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universidad Virgen Del Rocio, Seville
  - Hospital Mutua de Terrassa, Terrassa
  - Hospital Clinico Universitario de Valencia, Valencia
  - Unidad De Oncol/Hemat. Hospital, Valencia
  - Complexo Hospitalario Xeral de Vigo, Vigo Pontevedra
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza
- Karolinska University Hospital - Huddinge, Stockholm, Sweden
- Switzerland (2):
  - Kantonsspital Bruderholz, Bruderholz
  - UniversitaetsSpital Zuerich, Zurich
- Ibn-i Sina Hospital, Ankara, Turkey (Türkiye)
- United Kingdom (39):
  - Stoke Mandeville Hospital, Aylesbury-Buckinghamshire, England
  - Royal United Hospital, Bath, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Royal Bournemouth Hospital, Bournemouth, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Huddersfield Royal Infirmary, Huddersfield, West Yorks, England
  - Hull Royal Infirmary, Hull, England
  - Kettering General Hosptial, Kettering, Northants, England
  - Clinical Trials and Research Unit of the University of Leeds, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool and Broadgreen Hospitals NHS Trust, Liverpool, England
  - Liverpool University Hospital, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - St. Thomas' Hospital, London, England
  - Clinique Sainte Elisabeth, London, England
  - St. Georges, University of London, London, England
  - University College Hospital - London, London, England
  - Middlesex Hospital, London, England
  - James Paget Hospital, Norfolk, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Pontefract General Infirmary, Pontefract West Yorkshire, England
  - Rotherham District General Hospital - NHS Trust, Rotherham, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Southampton University Hospital NHS Trust, Southampton, England
  - Staffordshire General Hospital, Stafford, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Princess Margaret Hospital, Swindon, England
  - Hillingdon Hospital, Uxbridge, England
  - Sandwell General Hospital, West Bromwich, England
  - Centre for Cancer Research and Cell Biology at Belfast City Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland
  - Pinderfields Hospital NHS Trust, Wakefield, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Prince Philip Hospital, Dyfed, Wales
  - Singleton Hospital of the Swansea NHS Trust, Swansea, Wales

REFERENCES:
- [Derived] Pettengell R, Schmitz N, Gisselbrecht C, Smith G, Patton WN, Metzner B, Caballero D, Tilly H, Walewski JA, Bence-Bruckler I, To B, Geisler CH, Schots R, Kimby E, Taverna CJ, Kozak T, Dreger P, Uddin R, Ruiz de Elvira C, Goldstone AH. Rituximab purging and/or maintenance in patients undergoing autologous transplantation for relapsed follicular lymphoma: a prospective randomized trial from the lymphoma working party of the European group for blood and marrow transplantation. J Clin Oncol. 2013 May 1;31(13):1624-30. doi: 10.1200/JCO.2012.47.1862. Epub 2013 Apr 1. PMID 23547078